CLINICAL TRIAL: NCT03315039
Title: Phase 1/2 Study of Liposomal Annamycin for the Treatment of Subjects With Acute Myeloid Leukemia (AML) That is Refractory to or Relapsed After Standard Induction Therapy
Brief Title: Study of Liposomal Annamycin for the Treatment of Subjects With Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Moleculin Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MB-104
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Results first posted 2022-02-23 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Liposomal annamycin (Experimental): 2-hour intravenous infusion liposomal annamycin daily for 3 consecutive days followed by 18 days off study drug (i.e., one treatment cycle = 21 days).
  Interventions: Drug: Liposomal Annamycin

INTERVENTIONS:
Drug: Liposomal Annamycin — 2-hour intravenous infusion liposomal annamycin daily for 3 consecutive days followed by 18 days off study drug (i.e., one treatment cycle = 21 days).

SUMMARY:
This is a multi-center, open-label, dose escalation study that will determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of liposomal annamycin as a single agent for the treatment of subjects with AML that is refractory to or relapsed after standard induction therapy

ELIGIBILITY:
Inclusion Criteria:

1. A pathologically confirmed diagnosis of AML by World Health Organization (WHO) classification.
2. AML that is refractory to or relapsed after standard induction therapy.
3. Age ≥18 years at the time of signing informed consent.
4. No chemotherapy, radiation, or major surgery within two weeks prior to first dose of study drug and/or recovered from the toxic side effects of that therapy, unless treatment is indicated due to progressive disease.
5. No investigational therapy within four weeks of the first dose of study drug.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
7. Adequate laboratory results including the following:

   1. Bilirubin ≤1.5 times the upper limit of normal (ULN) unless due to Gilbert Syndrome
   2. Serum glutamic-oxaloacetic transaminase (SGOT), serum glutamic-pyruvic transaminase (SGPT) and alkaline phosphatase <3 times the ULN) unless due to organ involvement
   3. Adequate renal function (The Cockcroft-Gault equation will be used to estimate creatinine clearance. This equation is as follows: Creatinine clearance in ml/min = (140 - age) x body weight (kg)/72 x plasma creatinine (mg/dL); multiplied by 0.85 for women. Using this equation, adequate renal function will be deemed to be a creatinine clearance of greater than 60 ml/minute.)
8. Prior anthracycline cumulative dose below 551 mg/m2 or the daunorubicin equivalent which is the recommended non-cardiotoxic level.
9. Subject can understand and sign the informed consent document, can communicate with the investigator, and can understand and comply with the requirements of the protocol.
10. Women of childbearing potential must have a negative serum or urine pregnancy test.
11. All men and women must agree to practice effective contraception during the entire study period and after discontinuing study drug, unless documentation of infertility exists.

    1. Sexually active, fertile women must use two effective forms of contraception (abstinence, intrauterine device, oral contraceptive, or double barrier device) from the time of informed consent and until at least 6 months after discontinuing study drug
    2. Sexually active men and their sexual partners must use effective contraceptive methods from the time of subject informed consent and until at least 3 months after discontinuing study drug

Exclusion Criteria:

1. Subjects diagnosed with Acute Promyelocytic Leukemia.
2. Concomitant therapy that includes other chemotherapy that is or may be active against AML except for prophylaxis and/or treatment of opportunistic or other infection with antibiotics, antifungals and/or antiviral agents.
3. Prior mediastinal radiotherapy
4. Any condition which, in the opinion of the Investigator, places the subject at unacceptable risk if he/she were to participate in the study.
5. Positive risk assessment for cardiovascular disease including prior anthracycline cumulative dose more than 50% above recommended non-cardiotoxic levels, left ventricular ejection fraction (LVEF) <50%, valvular heart disease, or severe hypertension, (see Table 1). Cardiac subjects with a New York Heart Association (NYHA) classification of 3 or 4 will be excluded. (Cardiology consultation should be requested if any question arises about cardiac function.) This also includes subjects with baseline QT/QTc interval >480 msec, a history of additional risk factors for TdP (e.g., heart failure, hypokalemia, family history of Long QT Syndrome) and using concomitant medications that significantly prolong the QT/QTc interval.
6. Clinically relevant serious co-morbid medical conditions including, but not limited to, active infection, recent (less than or equal to six months) myocardial infarction, unstable angina, symptomatic congestive heart failure, uncontrolled hypertension, uncontrolled cardiac arrhythmias, chronic obstructive or chronic restrictive pulmonary disease, active CNS disease uncontrolled by standard of care, known positive status for human immunodeficiency virus (HIV) and/or active hepatitis B or C, cirrhosis, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Pregnant, lactating, or not using adequate contraception.
8. Known allergy to anthracyclines.
9. Any evidence of mucositis/stomatitis or previous history of severe (≥Grade 3) mucositis from prior therapy.
10. Required use of strong inhibitors and inducers of CYP enzymes and transporters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Shepard, MD, Study Director — Moleculin Biotech, Inc.
Locations (4):
- United States (4):
  - UC San Diego Health, La Jolla, California
  - University of Florida, Gainesville, Florida
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Southwest Cancer Center, Lubbock, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: no participants were enrolled in Phase 2
Groups:
- Dose Level 1: 100 mg/m2/Day Liposomal Annamycin; Dose Level 2: 120 mg/m2/Day Liposomal Annamycin: Liposomal Annamycin: 2-hour intravenous infusion liposomal annamycin daily for 3 consecutive days followed by 18 days off study drug (i.e., one treatment cycle = 21 days).
Period: Overall Study
Arm/Group | Dose Level 1: 100 mg/m2/Day Liposomal Annamycin | Dose Level 2: 120 mg/m2/Day Liposomal Annamycin
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1: 100 mg/m2/Day Liposomal Annamycin | Dose Level 2: 120 mg/m2/Day Liposomal Annamycin | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (6.73) | 57.0 (18.19) | 62.7 (12.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 3 | 7
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG grading scale- 0 - Fully active, able to carry on all pre-disease performance without restriction
  1- Restricted in physically strenuous activity but ambulatory and able to carry out work of a light of sedentary nature, e.g., light house work, office work 2 - Ambulatory and capable of all self care but unable to carry out any work activities. Up and about more than 50% of waking hours 3 - Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours 4 - Completely disabled. Cannot carry on any self care. Totally confined to bed or chair.
  5 - Dead
  Participants
    ECOG - 0 | 0 | 1 | 1
    ECOG - 1 | 3 | 1 | 4
    ECOG- 2 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicity
Description: Number of patients with a dose-limiting toxicity (DLT) at each dose evaluated
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 2 : 120 mg/m2/Day Liposomal Annamycin: Liposomal Annamycin: 2-hour intravenous infusion liposomal annamycin daily for 3 consecutive days followed by 18 days off study drug (i.e., one treatment cycle = 21 days).
Arm/Group | Dose Level 1: 100 mg/m2/Day Liposomal Annamycin | Dose Level 2 : 120 mg/m2/Day Liposomal Annamycin
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0

2. Secondary Outcome: Pharmacokinetics - Area Under the Plasma Concentration
Description: Area under the plasma concentration - time curve (AUC) of annamycin and its metabolite, annamycinol
Time Frame: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, and 24 hours after the start of liposomal annamycin infusion on Day 1 and Day 3
Population: One participant excluded from summary statistics due to high Annamycin concentrations
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/ml
Arm/Group | Liposomal Annamycin
Number analyzed (Participants) | 6
hr*ng/ml
  Annamycin 100 mg/m2 - Day 1: number analyzed (Participants) | 4
  Annamycin 100 mg/m2 - Day 1 | 1430 (19.6)
  Annamycin 100 mg/m2 - Day 3: number analyzed (Participants) | 4
  Annamycin 100 mg/m2 - Day 3 | 1610 (22.4)
  Annamycin 120 mg/m2 - Day 1: number analyzed (Participants) | 2
  Annamycin 120 mg/m2 - Day 1 | 2330 (42.0)
  Annamycin 120 mg/m2 - Day 3: number analyzed (Participants) | 2
  Annamycin 120 mg/m2 - Day 3 | 2880 (33.3)
  Annamycinol 100 mg/m2 - Day 1: number analyzed (Participants) | 4
  Annamycinol 100 mg/m2 - Day 1 | 1400 (43.9)
  Annamycinol 100 mg/m2 - Day 3: number analyzed (Participants) | 4
  Annamycinol 100 mg/m2 - Day 3 | 1520 (36.7)
  Annamycinol 120 mg/m2 - Day 1: number analyzed (Participants) | 2
  Annamycinol 120 mg/m2 - Day 1 | 1370 (39.5)
  Annamycinol 120 mg/m2 - Day 3: number analyzed (Participants) | 2
  Annamycinol 120 mg/m2 - Day 3 | 1610 (67.7)

3. Secondary Outcome: Number of Participants With Anti-leukemic Activity
Description: Determined by acute myeloid leukemia (AML) response rate based on the International Working Group (IWG) Response Criteria in AML (Cheson, 2003). Anti-leukemic Activity measured by bone marrow biopsy/aspirate pre and post treatment.
Time Frame: 15-35 Days after the start of therapy
Measure: Count of Participants; unit: Participants
Groups:
- 100 mg/m2: Best Overall Response for Participants treated at 100 mg/m2 dose level
- 120 mg/m2: Best Overall Response for treated at 120 mg/m2 dose level
Arm/Group | 100 mg/m2 | 120 mg/m2
Number analyzed (Participants) | 4 | 3
Participants
  Morphological Leukemia Free State (MLFS) | 0 | 1
  Treatment Failure (TF) | 4 | 2

ADVERSE EVENTS:
Time Frame: 39 days after the last dose of study treatment, a total of about 1 year and 10 months since the start of the study.
Description: AEs were collected from safety population from the time of study treatment initiation until 39 days after the last dose of study treatment.
  Safety population = all participants who received any amount of liposomal annamycin.
Groups:
- 100 mg/m2 Dose Level; 120 mg/m2 Dose Level: Liposomal Annamycin: 2-hour intravenous infusion liposomal annamycin daily for 3 consecutive days followed by 18 days off study drug (i.e., one treatment cycle = 21 days).
Arm/Group | 100 mg/m2 Dose Level | 120 mg/m2 Dose Level
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 100 mg/m2 Dose Level (N=4) | 120 mg/m2 Dose Level (N=3)
Flank Pain (General disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 100 mg/m2 Dose Level (N=4) | 120 mg/m2 Dose Level (N=3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Lip Dry (Gastrointestinal disorders) | 0 | 1
Oral Pain (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Platelet count decreased (Investigations) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
White blood cell count decreased (Investigations) | 2 | 1
Blood creatinine increased (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Asparate aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1
Weight Increased (Investigations) | 0 | 1
Decreased apetite (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1
Fluid Overload (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Pain of Skin (Skin and subcutaneous tissue disorders) | 0 | 1
Visual impairment (Eye disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 1
Escherichia bacteraemia (Infections and infestations) | 1 | 1
Folliculitis (Infections and infestations) | 2 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Enterococcal infection (Infections and infestations) | 0 | 1
Pneumonia fungal (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Skin Wound (Injury, poisoning and procedural complications) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Mucosal iflammation (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Urinary hesitation (Renal and urinary disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT03315039/Prot_SAP_001.pdf